CLINICAL TRIAL: NCT07273578
Title: Home Blood Pressure Monitoring in Patients With Uncontrolled Hypertension: a Randomized Clinical Trial
Acronym: HP-HBMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Ceara (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Antonia Fabiana Rodrigues da Silva, Doutora, Universidade Federal do Ceara
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: nº 5.769.427
Record Dates: First submitted 2025-01-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure Determination; UNCONTROLLED HYPERTENSION
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The intervention consisted of implementing HBPM to individuals with uncontrolled hypertension who were allocated to the IG, where they performed four measurements per day, two in the morning and two at night, before meals, for 5 consecutive days each month during follow-up, during three follow-up appointments at the unit. They also received a monthly telephone call to remind them to perform the measurements.
Who Masked: Outcomes Assessor
Masking Description: The final data was anonymized before being made available to the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grupo intervenção (GI) (Active Comparator): The intervention consisted of HBPM being performed by IG participants, who were loaned an automatic BP monitor to take measurements at home, for 5 consecutive days each month.
  Interventions: Procedure: Home Blood Pressure Monitoring
- Grupo controle (GC) (No Intervention)

INTERVENTIONS:
Procedure: Home Blood Pressure Monitoring — The intervention consisted of HBPM being performed by IG participants, who were loaned an automatic BP monitor to take measurements at home, for 5 consecutive days each month.
  Arms: Grupo intervenção (GI)

SUMMARY:
This study aimed to test Home Blood Pressure Monitoring (HBPM) in reducing blood pressure (BP) levels in individuals with uncontrolled hypertension. Data collection was conducted in 5 stages: 1) recruitment; 2) inclusion in the study and collection of baseline data, including information on sociodemographic issues, anthropometric and clinical profile, and adherence to medication treatment; 3) randomization; 4) intervention; and 5) Reassessment of adherence to medication treatment. All participants will be monitored by the research team in three follow-up visits at the unit. The intervention consisted of HBPM being performed by participants in the IG, who were loaned an automatic BP monitor to take measurements at home, for 5 consecutive days each month. Participants in the CG did not perform HBPM, but were also monitored by the research team in their follow-up visits. In these follow-up visits, for both groups, the researchers performed new BP measurements using the oscillometric method.

DETAILED DESCRIPTION:
The outcome was the reduction in mean SBP and DBP values over time within and between groups, consisting of a reduction with a significant difference between the baseline and the post-intervention period.

The Omron HEM-1100® automatic clinical monitor was used to perform oscillometric BP measurement in the unit.

The HEM 7122 automatic BP monitor was made available to IG participants for self-measurement of BP at home. The following were included:

1. Patients diagnosed with hypertension associated or not with DM, CAD or RI;
2. Time since diagnosis greater than 6 months;
3. BP > 140/90 mmHg obtained in triplicate during an initial clinical consultation conducted by the researchers, immediately after the invitation to participate in the study;
4. They had been following the same antihypertensive drug treatment for at least 4 weeks, according to the participant's self-report;
5. They were able to move around and attend follow-up appointments at the health unit. The random allocation of participants into the two groups (G1 and CG) was performed proportionally (1:1) using Research Randomizer 1, which generated the sequence of entry by sets (set 01: G1, Set 02: CG). The numbers generated were previously recorded in sealed envelopes, which were opened in the presence of the participants immediately after collecting the variables at baseline and completing the data collection instrument. After randomization, the researcher informed the IG participant that he would undergo the intervention with HBPM during the follow-up period of three consecutive appointments scheduled by the unit. To this end, he would be loaned an automatic BP monitor provided by the researcher for the duration of the study and that it should be returned at the end. The CG participant was also informed by the researcher about the monitoring by the research team, which would include taking BP measurements using the oscillometric method during the period of three consecutive return appointments scheduled by the unit.

ELIGIBILITY:
Inclusion criteria: a) Patients diagnosed with hypertension, whether or not associated with DM, CAD or RI; b) Time since diagnosis greater than 6 months; c) BP > 140/90 mmHg obtained in triplicate during the initial clinical consultation conducted by the researchers, immediately after the invitation to participate in the study; d) Having been following the same antihypertensive drug treatment for at least 4 weeks, according to the participant's self-report; e) Having mobility conditions to attend follow-up consultations at the health unit.

Exclusion Criteria: a) Pregnant women or women actively seeking to become pregnant; b) Have physical incapacity (represented by the presence of tetraplegia, tetraparesis, triplegia, triparesis, hemiplegia, hemiparesis, amputation or cerebral palsy), cognitive incapacity (represented by the presence of dementia, depression, delirium and mental illnesses, such as schizophrenia, oligophrenia and paraphrenia), and have undergone surgical procedures, accidents, amputation, oncological treatment that prevents self-monitoring of BP; c) Inability to maintain the monitor at home, represented by the participant's refusal to receive and/or keep the device; d) Acute cardiovascular event (myocardial infarction and stroke) in the last three months; e) Have a medical diagnosis of arrhythmia, as per the participant's self-report and confirmation in the medical record. f) Perform home BP measurement, represented by the participant's report. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Reduction in average Systolic and Diastolic Blood Pressure values | 9 months
  Reduction in mean SBP and DBP values over time within and between groups, consisting of a reduction with a significant difference between the baseline and the post-intervention period.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal do Ceará, Fortaleza, Ceará/BRASIL, Brazil

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: Data de inicio ainda não foi prevista
Access Criteria: Those who request